CLINICAL TRIAL: NCT05016063
Title: Phase I Study to Evaluate the Safety and Effectiveness of Dual CD33-CLL1 CAR-T Therapy in Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Dual CD33-CLL1-CAR-T Cells in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xi Zhang, MD, Chef of Hematology Department, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dual CD33-CLL1 CAR-T cells
Record Dates: First submitted 2021-08-14; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual CD33-CLL1 CAR-T cells (Experimental): CD33-CLL1 CAR T cells
  Interventions: Drug: Fludarabine; Drug: Cytoxan; Biological: Dual CD33-CLL1 CAR-T cells

INTERVENTIONS:
Drug: Fludarabine — recommendation: 30mg/m2 (D-5~D-3),determined by tumor burden at baseline.
Drug: Cytoxan — recommendation: 300-500mg/m2 (D-5~D-3),determined by tumor burden at baseline.
Biological: Dual CD33-CLL1 CAR-T cells — CD33-CLL1 CAR-T infusion (starting at dose level 1 [DL1]: 0.5 x 106 transduced CAR-T cells/kg) on Day 0.

SUMMARY:
Phase I, interventional, single-arm, open-label, treatment study to evaluate the safety and effectiveness of CD33-CLL1 CAR in patients with relapsed and/or refractory acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
AML bears heterogeneous cells that can consequently offset killing by single-CAR-based therapy, which results in disease relapse. Leukemic stem cells (LSCs) associated with CLL1 expression comprise a rare population that also plays an important role in disease progression and relapse for myeloid malignancies. CD33 is widely expressed in AML. Targeting both CD33 and CLL1 surface antigens together may offer two distinct benefits. First, targeting both bulk disease and leukemic stem cells together allows for a more comprehensive ablation of the disease. Second, dual targeting of myeloid malignancies by both CD33 and CLL1 directed therapy overcomes the pitfalls of single-antigen therapy by preventing relapse due to antigen loss. While loss of a single antigen under antigen-specific selection pressure is possible, loss of two antigens simultaneously is much less likely.

CD33-CLL1 CAR is a compound Chimeric Antigen Receptor immunotherapy with two distinct functional CAR molecules expressed on a T-cell, directed against the surface proteins CLL1 and CD33. CD33-CLL1 CAR intends to target the mechanisms of single-CAR relapse, specifically antigen escape and leukemic stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status score ≤ 2.
2. Life expectancy ≥ 12 weeks from the time of enrollment.
3. Disease status at the time of enrollment: -Patients with AML (except M3) who have not achieved complete remission after standard chemotherapy regimens; -Not suitable or unconditional for allogeneic hematopoietic stem cell transplantation; -Patients with recurrent acute myeloid leukemia after autologous hematopoietic stem cell transplantation without active graft-versus-host disease (GVHD).
4. CD33 expression must be detected on greater than 50% of the malignant cells by immunohistochemistry or greater than 80% by flow cytometry.
5. Adequate main organ function as assessed by the following laboratory requirements: creatinine ≤ 2.5 × upper limit of normal, cardiac ejection fraction ≥ 40%, oxygen saturation ≥ 90%, total bilirubin ≤ 3 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, Hgb≥80g/L.
6. Without history of accepting anti-cancer therapy, including chemotherapy, radiotherapy, immunotherapy (immune suppressive drugs or corticosteroid treatment) within 4 weeks of screening.
7. Women of child-bearing age must have evidence of negative pregnancy test.
8. Subjects of reproductive potential must agree to use acceptable birth control methods within 1 year after treatment, as described in protocol.
9. After discussion by the expert group, the patient's condition was analyzed and combined with the general physical condition of the patient, the benefit of participating in the clinical trial was greater than the risk.
10. All participants must have the ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL M3): t(15;17)(q22;q12); (promyelocytic leukemia [PML]/retinoic acid receptor [RAR] alpha [a]) and variants excluded.
2. Active acute or chronic GVHD or requirement of immunosuppressant medications for GVHD within 4 weeks of enrollment.
3. Have been diagnosed with or treated other malignant tumors other than AML within 5 years before screening, except for the following conditions: participants with adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer; or received radical treatment Local prostate cancer, ductal carcinoma in situ.
4. There are serious systemic diseases: New York Heart Association (NYHA) stage III or IV congestive heart failure; cerebrovascular accident or myocardial infarction or hemodynamic instability caused by arrhythmia within 6 months before signing the informed consent; impaired cardiac function (LVEF<50%) assessed by echocardiographic scan.
5. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
6. Pregnant or lactating women.
7. Subjects with radiologically-detected CNS chloromas or CNS 3 disease (presence of ≥ 5/μL white blood cells (WBCs) in cerebral spinal fluid (CSF) and cytospin positive for blasts [in the absence of a traumatic lumbar puncture] and/or clinical signs of CNS leukemia such as a cranial nerve palsy from active disease). Subjects with adequately treated CNS leukemia are eligible.
8. Human immunodeficiency virus (HIV) seropositivity; hepatitis B surface antigen is positive or HBV DNA is higher than the detection limit of the analysis method; hepatitis C antibody is positive or HCV RNA is higher than the detection limit of the analysis method; syphilis antibody and syphilis rapid plasma reagin are positive; CMV DNA is positive.
9. Patients who suffer from allergies for any cytokines or antibodies.
10. Contraindications for fludarabine or cyclophosphamide treatment.
11. Receiving corticosteroids at >20 mg daily prednisone dose or equivalent.
12. Drug abuse and addiction.
13. History of mental disorders.
14. Other patients that researchers considered unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 4 weeks after infusion
  Assessment of morphologic complete remission (CR), complete remission with incomplete recovery of counts (CRi), no residual disease as analyzed by flow cytometry analysis, and molecular remission by molecular studies
the safety evaluation of Dual CD33-CLL1 CAR-T cells | within 4 weeks after infusion
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years after infusion
  Surviavl without disease progression
Overall survival(OS) | up to 2 years after infusion
  Surviavl

CONTACTS AND LOCATIONS:
Overall Officials: xi zhang, PhD/MD, Principal Investigator — Department of Hematology, Xinqiao Hospital
Locations (1):
- Department of Hematology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No